CLINICAL TRIAL: NCT06405308
Title: Robotic Natural Orifice Specimen Extraction Surgery Versus Robotic Transabdominal Specimen Extraction Surgery for Rectal Cancer: a Multicentre Propensity Score-Matched Analysis
Brief Title: Robotic Natural Orifice Specimen Extraction Surgery Versus Robotic Transabdominal Specimen Extraction Surgery for Early-Stage Rectal Cancer
Status: Completed | Type: Observational
Sponsor: Taiyuan Li (Other)
Responsible Party: Sponsor-Investigator, Taiyuan Li, Professor, The First Affiliated Hospital of Nanchang University
Organization: The First Affiliated Hospital of Nanchang University (Other)
Other Study IDs: NOSES-2024
Record Dates: First submitted 2024-05-04; First posted 2024-05-08 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Rectal Cancer; Robotic Surgery; Natural Orifice Specimen Extraction Surgery
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- R-NOSES group: Participants in this group underwent robotic natural orifice specimen extraction surgery
  Interventions: Procedure: R-NOSES group
- R-TSES group: Participants in this group underwent robotic transabdominal specimen extraction surgery
  Interventions: Procedure: R-TSES group

INTERVENTIONS:
Procedure: R-NOSES group — robotic natural orifice specimen extraction surgery
  Groups: R-NOSES group
Procedure: R-TSES group — robotic transabdominal specimen extraction surgery
  Groups: R-TSES group

SUMMARY:
A retrospective cohort study, conducted nationwide（China） and across multiple centers, aimed to compare the surgical quality and short-term outcomes of R-NOSES （robotic natural orifice specimen extraction surgery）with R-TSES （robotic transabdominal specimen extraction surgery） for early-stage rectal cancer.

DETAILED DESCRIPTION:
In this retrospective cohort study, data from 1086 patients who underwent R-NOSES or R-TSES for early-stage rectal cancer between October 2015 and November 2023 were collected from a prospectively maintained database of 8 experienced surgeons from 8 high-volume centers in china. The study was aimed to compare the surgical quality and short-term outcomes of R-NOSES with R-TSES for early-stage rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. histologically confirmed rectal adenocarcinoma
2. robotic TME for rectal adenocarcinoma
3. postoperative pathological staging of T1-2N0M0
4. complete surgical and postoperative follow-up information

Exclusion Criteria:

1. body mass index (BMI) ≥ 35 kg/m2
2. history of abdominal surgery
3. history of pelvic surgery
4. presence of another primary cancer
5. previous endoscopic submucosal dissection (ESD) or endoscopic mucosal resection (EMR)
6. anal or vaginal disease
7. ileostomy or transverse colostomy
8. conversion to open operation
9. tumor distant metastasis

Ages: 20 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent R-NOSES or R-TSES for early-stage rectal cancer between October 2015 and November 2023.
Sampling Method: Non-Probability Sample
Enrollment: 636 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Complication rate | Up to 30 days postoperatively
  Complication rate within 1 month postoperatively.All complications of surgery will be documented and graded by the Clavien-Dindo classification system,generally including anastomotic leakage, abdominal infection, bleeding, incision infection, incision implantation, intestinal obstruction, and rectovaginal fistula.

SECONDARY OUTCOMES:
Operative time | Intraoperative
Estimated blood loss | Intraoperative
Postoperative recovery composite | Up to 2 weeks
  Including the time to first flatus (record the patient's first self induced exhaust time after operation, accurate to hours) and time to first oral feeding.
Postoperative hospital stay | Up to 4 weeks
  From surgery to discharge
Pain assessment | 1, 3, 5 days postoperatively
  Visual analogue scale (VAS) will be used to evaluate the postoperative pain. If analgesics were needed, the type and dose of analgesics after operation should be recorded.
C-reactive protein (CRP) | 1, 3, 5 days postoperatively
  Detection of serum CRP levels (mg/L) to evaluate surgical stress response and immune function.
Postoperative white blood | 1, 3, 5 days postoperatively
  Detection of serum CRP levels (mg/L) to evaluate surgical stress response and immune function.
EORTC QLQ-C30 | Three months after surgery
  The EORTC QLQ-C30 includes functional score, symptom score, and Global Health Status. All project scores range from 0 to 100. The Functional score includes physical functioning, role functioning, emotion functioning, social functioning and cognitive functioning. The higher the functional score, the better the functional status of the patient. Symptom score includes nausea and vomiting, pain, dyspnoea, insomnia, loss of appetite, constipation, diarrhea, financial impact. A higher symptom score is associated with more severe symptoms and worse outcomes. The higher the Global Health Status, the better the health of the patient.
BIQ | Three months after surgery
  The BIQ is an eight-item questionnaire incorporating body image and cosmetic subscales, The body image scale measures patients' perception and satisfaction with their bodies after surgery. it ranges from 5 to 20 with a higher number representing greater body image perception. The cosmetic scale assesses satisfaction with surgical scars for a score range of 3-24, with a higher score indicating greater cosmetic satisfaction.

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing
  - Three Gorges Hospital Affiliated to Chongqing University, Chongqing
  - Fujian Cancer Hospital, Fuzhou
  - The Second Affiliated Hospital of Harbin Medical University, Harbin
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Zhongshan Hospital, Fudan University, Shanghai
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou